CLINICAL TRIAL: NCT04987658
Title: A Phase 1, Multiple-dose, Open-label Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of OLZ/SAM in Pediatric Subjects (10-12 Years Old) With Bipolar I Disorder
Brief Title: Phase 1 Study of OLZ/SAM in Pediatric Subjects With Bipolar I Disorder
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alkermes, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ALKS 3831-A311
Record Dates: First submitted 2021-07-26; First posted 2021-08-03 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Bipolar I Disorder
Keywords: Bipolar I Disorder; Olanzapine; Samidorphan; OLZ/SAM; ALKS 3831; Pediatric pharmacokentics; LYBALVI

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group 1 Olanzapine/ 5 mg Samidorphan (Experimental): Olanzapine will be gradually increased to a target dose of 10mg/samidorphan 5mg (Range: 5-20mg Olanzapine/samidorphan 5mg)
  Interventions: Drug: OLZ/SAM
- Group 2 Olanzapine/ 10mg Samidorphan (Experimental): Olanzapine will be gradually increased to a target dose of 10mg/samidorphan 10mg (Range: 5-20mg Olanzapine/samidorphan 10mg)
  Interventions: Drug: OLZ/SAM

INTERVENTIONS:
Drug: OLZ/SAM — Olanzapine and Samidorphan taken once daily over a max period of 21 days
  Other Names: ALKS 3831

SUMMARY:
To evaluate the safety, tolerability, and pharmacokinetics of olanzapine and samidorphan in clinically stable pediatric subjects (10 to 12 years old) with Bipolar I disorder following oral administration of multiple ascending doses of OLZ/SAM

ELIGIBILITY:
Inclusion Criteria:

* Subject's parent(s)/legal guardian(s) is considered reliable by the Investigator and has agreed to provide support to the subject to ensure compliance with study treatment, visits, and protocol procedures.
* Male and female subjects between 10 and 12 years of age, inclusive.
* Subject weighs ≥70 pounds.
* Subjects who are receiving antipsychotic treatment for their medical condition, with a diagnosis of bipolar I disorder.
* Subjects must be considered stable, per investigator judgement.
* Subject is willing to abide by the contraception requirements for the duration of the study.

Exclusion Criteria:

* Subject has a comorbid neuropsychiatric disorder that could interfere with participation in the study.
* Subject poses a current suicide risk as assessed by the Investigator or as confirmed by the baseline Columbia-Suicide Severity Rating Scale by a response of "Yes" to question numbers 4 or 5 with ideation or suicidal behavior occurring in the past 12 months (assessed at Screening and at Visit 2, Day 1).
* Subject has a diagnosis of diabetes or presents with pre-diabetes lab results (hemoglobin A1c ≥6%).
* Subject has a history of use of clozapine or use of long-acting injectable antipsychotic medication within 3 months prior to Screening.
* Subject has a DSM-5 (Diagnostic and Statistical Manual of Mental Disorders-5) diagnosis of moderate to severe alcohol disorder, or moderate to severe substance use disorder, within the 3 months prior to Screening.
* Subject has taken opioid agonists within the 14 days prior to Screening, or has taken long-acting opioid agonist within the 30 days prior to Screening, or has anticipated a need to take opioid medication during the study period (eg, planned surgery, including oral surgery), or has taken opioid antagonists including naltrexone (any formulation) and naloxone within 60 days prior to Screening.
* Subject is unable to swallow oral medications, as assessed by the Investigator.
* Subject has a positive urine drug screen for opioids (assessed at Screening and at Visit 2, Day 1).
* Subject has a positive cotinine test (assessed at Screening and at Visit 2, Day 1).
* Subject has an intellectual disability, as assessed by the Investigator.
* Subject has a history of intolerance or hypersensitivity to olanzapine or opioid antagonists, or any component of the study drug.

Ages: 10 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 7 (Actual)
Dates: Start 2021-07-22 (Actual); Primary Completion 2023-08-11 (Actual); Study Completion 2023-08-11 (Actual)

PRIMARY OUTCOMES:
Maximum plasma concentration observed | Up to 3 weeks
Area under the plasma concentration-time curve over the 24-hour dosing interval | Up to 3 weeks
Time to reach maximum concentration | Up to 3 weeks
Incidence of Adverse Events | Up to 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: David McDonnell, MD, Study Director — Alkermes, Inc.
Locations (2):
- United States (2):
  - Alkermes Investigational Site, Decatur, Georgia
  - Alkermes Clinical Investigative Site, Cincinnati, Ohio

IPD SHARING:
Plan to Share IPD: No